CLINICAL TRIAL: NCT02297594
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of AK0529 When Administered Orally in Healthy Male and Female Adult Subjects
Brief Title: Safety, Tolerability and PK Study of AK0529 in Healthy Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK0529-1001
Record Dates: First submitted 2014-11-11; First posted 2014-11-21 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — ziresovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AK0529 (Experimental): Generic name: AK0529 Dosage Form: capsule
  Interventions: Drug: AK0529
- Placebo (Placebo Comparator): Sugar placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK0529 — AK0529 capsule for oral administration
  Other Names: AK0529 capsule
  Arms: AK0529
Drug: Placebo — Sugar placebo capsule for oral administration
  Other Names: Sugar placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and PK of single and multiple ascending dose of AK0529 when administered orally in healthy subjects

DETAILED DESCRIPTION:
This is a Phase 1, first-in-man, single-center, randomized, double blind, placebo controlled single and multiple ascending dose study in healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Must be healthy males, or healthy females of non-childbearing potential or surgically sterilized or post-menopausal (amenorrhea for at least 1 year and confirmed by a follicle stimulating hormone [FSH] result of > 20 IU/mL).
2. Must be aged 18 to 55 years of age inclusive.
3. Must have body mass index (BMI) of 18.0 to 31.0 kg/m2 inclusive.
4. Must have total body weight ≥50 kg at screening but ≤100 Kg.
5. Must be willing and able to communicate and participate in the whole study.
6. Must provide written informed consent.
7. Must agree to use an adequate method of contraception (as defined in Section 4.2.1).
8. Must have AST, ALT, total bilirubin, urea, creatinine and hemoglobin within the laboratory reference range at screening and Day -1.
9. Must have QTcF <450 ms, QTcB <450 ms and PR interval <210 ms for screening, Day -1 and pre-dose ECG measurements, and not have any degree of heart block or conduction abnormality.
10. Must have serology demonstrating they are free from infection with hepatitis B, hepatitis C, and human immunodeficiency virus (HIV-1 and HIV-2)

Exclusion Criteria:

1. Male subjects who have currently pregnant partners or who have partners planning to become pregnant during the duration of the study.
2. Evidence or history of clinical significant oncological, pulmonary, chronic respiratory, hepatic, cardiovascular, hematological, metabolic, neurological, immunological, nephrological, endocrine or psychiatric disease, or current infection.
3. Clinically relevant (as decided by the investigator and the medical monitor) abnormalities in the ECG (12 standard leads) including any degree of heart block, including asymptomatic bundle branch block.
4. Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
5. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
6. Electrolyte disturbances, particularly hypokalemia hypocalcemia or hypomagnesemia.
7. Any condition that could possibly affect drug absorption, e.g. gastrectomy or diarrhea.
8. History of post-antibiotic colitis.
9. History of any drug or alcohol abuse in the past 2 years prior to screening.
10. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = 400 mL beer, 25 mL of 40% spirit or a 75 mL glass of wine).
11. Subjects who have a urine cotinine greater than 500 ng/mL at screening will be excluded. Subjects who are tobacco users (including smokers and users of snuff, chewing tobacco and other nicotine or nicotine-containing products) must have stopped use at least 90 days before screening.
12. Receipt of an investigational drug or participation in another clinical research study within 90 days prior to drug administration.
13. Subjects who are study site employees, or immediate family members of a study site or sponsor employee.
14. Subjects who have previously been enrolled and dosed in this study, except subjects undergoing repeat dosing in Cohort 4F (the fed PK cohort of the SAD part of the study).

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, serious adverse events | Screening to Day 14 - 21

SECONDARY OUTCOMES:
Pharmacokinetics of single dose study: Area Under Curve (AUC) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
Pharmacokinetics of single dose study: Observed Maximum plasma concentration (Cmax) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
Pharmacokinetics of single dose study: half-life (t1/2) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
Pharmacokinetics of single dose study: time to maximum plasma concentration (tmax) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
Pharmacokinetics of single dose study: Volume of distribution | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
Pharmacokinetics of single dose study: Clearance | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 and 48 hours post-dose
Pharmacokinetics of multiple dose study:Area Under Curve (AUC) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day1 and pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 hours post-dose on Day 7 and at 24 hours (Day 8) and at 48 hours (Day 9)
Pharmacokinetics of multiple dose study: Observed Maximum plasma concentration (Cmax) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day1 and pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 hours post-dose on Day 7 and at 24 hours (Day 8) and at 48 hours (Day 9)
Pharmacokinetics of multiple dose study: half-life (t1/2) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day1 and pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 hours post-dose on Day 7 and at 24 hours (Day 8) and at 48 hours (Day 9)
Pharmacokinetics of multiple dose study: time to maximum plasma concentration (tmax) | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day1 and pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 hours post-dose on Day 7 and at 24 hours (Day 8) and at 48 hours (Day 9)
Pharmacokinetics of multiple dose study:Volume of distribution | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day1 and pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 hours post-dose on Day 7 and at 24 hours (Day 8) and at 48 hours (Day 9)
Pharmacokinetics of multiple dose study: clearance | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8 and 12 hours post-dose on Day1 and pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 hours post-dose on Day 7 and at 24 hours (Day 8) and at 48 hours (Day 9)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffin, MD, Principal Investigator — Q-Pharm Pty Ltd
Locations (1):
- Q-Pharm Pty Ltd QIMR Berghofer & Royal Brisbane and Women's Hospital Campus, Brisbane, Queensland, Australia